CLINICAL TRIAL: NCT04151745
Title: Effect of Atrial Pacing on Right Ventricular Function After Cardiac Surgery
Acronym: Outpace
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: interaction with another study, not possible to include patients
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Principal Investigator, Frisius Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TPO
Record Dates: First submitted 2019-01-15; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Right Ventricular Ejection Fraction

STUDY DESIGN:
Intervention Model Description: To investigate the effects of atrial pacing on right ventricular function and hemodynamics after open heart surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): When a hemodynamically stable state is achieved, the external pacemaker will be switched off for 30 minutes. Hemodynamic parameters will be acquired directly prior to switching off, 15 respectively 30 minutes after switching off, and 15 minutes after switching back on. To gain insight in the natural course of stunning, this routine will be repeated the next morning.
  Interventions: Procedure: external pacemaker switched off

INTERVENTIONS:
Procedure: external pacemaker switched off — When a hemodynamically stable state is achieved, the external pacemaker will be switched off for 30 minutes. Hemodynamic parameters will be acquired directly prior to switching off, 15 respectively 30 minutes after switching off, and 15 minutes after switching back on. To gain insight in the natural course of stunning, this routine will be repeated the next morning.

SUMMARY:
Temporary pacing with an external pacemaker after open heart surgery - besides preventing arrhythmias and AV-conduction disorders - is used to improve cardiac output. In theory, postoperative stunning temporarily limits stroke volume and SA-node dysfunction compromises an adequate compensatory rise in heartrate to ensure sufficient cardiac output. There is a lack of consensus regarding the use of this form of pacing. Protocols vary widely between hospitals. Moreover, the scientific base for this form of pacing mainly comprises studies dating back to the nineteen sixties and seventies. Major changes in (operating) techniques have taken place since then. Also, the role of the right ventricle in this context has not been studied specifically. The current study aims to investigate the effects of atrial pacing on right ventricular function specifically and hemodynamics in general, in today's postoperative setting. We hypothesize that a reduction in heart rate may lead to decreased right ventricular function.

DETAILED DESCRIPTION:
When a hemodynamically stable state is achieved, the external pacemaker will be switched off for 30 minutes. Hemodynamic parameters will be acquired directly prior to switching off, 15 respectively 30 minutes after switching off, and 15 minutes after switching back on. To gain insight in the natural course of stunning, this routine will be repeated the next morning. No additional hemodynamic interventions will be allowed in these periods.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* admitted to the ICU after onpump open heart surgery
* Swan Ganz thermodilurion catheter in situ

Exclusion Criteria:

* participation other trials
* off pump cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
right ventricular ejection fraction | 30 minutes after procedure
  difference in right ventricular function expressed in RVEF

CONTACTS AND LOCATIONS:
Overall Officials: E C Boerma, Dr, Principal Investigator — Intensive Care

IPD SHARING:
Plan to Share IPD: No